CLINICAL TRIAL: NCT01439295
Title: Urinary Ascorbyl Peroxide as an Early Biological Marker of Bronchopulmonary Dysplasia in Preterm Infants Less Than 33 Weeks of Gestation
Brief Title: Ascorbyl Peroxide Association With Bronchopulmonary Dysplasia
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Ibrahim Mohamed, Adjunct professor of peditarics, division of neonatology, St. Justine's Hospital
Other Study IDs: University of Montreal; CIHR246505 (Other Grant/Funding Number: Canadain Institute of Health Research (CIHR))
Record Dates: First submitted 2011-09-16; First posted 2011-09-23 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Ascorbyl peroxide; Bronchopulmonary dysplasia; Redox status; Necrotising entercolitis; Retinopathy of prematurity; Patent ductus arteriosus; Intraventricular hemorrhage; Periventricular leucomalacia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Ductus Arteriosus, Patent; Leukomalacia, Periventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sample (650 µl) Blood sample (500 µl)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm less than 33 weeks: This cohort will be composed of premature infants born before 33 weeks of gestational age, admitted to the neonatal intensive care unit at Sainte-Justine hospital and receiving parenteral nutrition (PN) during their first week of life.

SUMMARY:
Urinary ascorbyl peroxide level in the first week of life will be a good predictor of Bronchopulmonary dysplasia (BPD) in preterm infants less than 33 weeks of gestation.

DETAILED DESCRIPTION:
This study uses ascorbyl peroxide as representative of oxidative stress in premature infants on parenteral nutrition and aims to test the correlation of this metabolite and the different major neonatal outcomes 'mainly bronchopulmonary dysplasia).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 33 weeks of gestation<
* Admission to CHU Sainte-JUstien neonatal intensive care unit
* Receiving Parenteral nutrition during the first week of life
* Parental consent

Exclusion Criteria:

* Major congenital anomalies
* Sever perinatal asphyxia

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants less than 33 weeks of getation
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Bronchopulmonary Dysplasia | 4 Months
  To correlate the level of urinary Ascorbyl peroxide and BPD. Full diagnosis and classification (to mild, moderate or severe) is at 36 weeks of corrected age; so even for most premature infants (like 23 weeks of gestation) there will be a need for follow up for less than 4 month to have the final diagnosis at 36 weeks

SECONDARY OUTCOMES:
The redox status (in blood) | First week of life (week 1) and 36 semaines CA
  Testing the correlation between the urinary level of ascorbyl peroxide and the redox status in the blood at 5 to 7 days of life. Measuring the Redox potential at 36 weeks corrected age to investigate long term effect of early oxidative stress.
Major neonatal outcomes (NEC, ROP, PDA, IVH, PVL) | 4 Months
  These outcomes are the major neonatal outcomes for preterm infants, we would test the correlation between ascorbyl peroxide (as marker of oxidative stress) and like Necrotising enterocolotis (NEC), Retinopathy of prematurity (ROP),patent ductus arteriosis(PDA), intraventricular hemorrhage (IVH) and periventricular leucomalacia (PVL).

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Mohamed, Mb CHB, Principal Investigator — University of Montreal, Sainte Justine Hospital; Jean-claude Lavoie, PhD, Study Director — University of Montreal, Sainte-Justine hospital research center
Locations (1):
- University of Montreal, Sainte-Justine Hospital, Montreal, Quebec, Canada

REFERENCES:
- See also: Neonatal Exposure to Oxidants Induces Later in Life a Metabolic Response Associated to a Phenotype of Energy Deficiency in an Animal Model of Total Parenteral Nutrition — http://journals.lww.com/pedresearch/Fulltext/2010/09000/Neonatal_Exposure_to_Oxidants_Induces_Later_in.2.aspx
- See also: Admixture of a Multivitamin Preparation to Parenteral Nutrition: The Major Contributor to In Vitro Generation of Peroxides — http://www.pediatricsdigest.mobi/content/99/3/e6.full
- See also: Paradoxical Role of Ascorbic Acid and Riboflavin in Solutions of Total Parenteral Nutrition: Implication in Photoinduced Peroxide Generation — http://journals.lww.com/pedresearch/pages/articleviewer.aspx?year=1998&issue=05000&article=00007&type=abstract